CLINICAL TRIAL: NCT00199979
Title: Multicenter, Randomized, Open-Label Trial, Assessing the Efficacy of Zidovudine, Lamivudine and Nevirapine Combination Administered Twice Daily, Versus the Association of Tenofovir, Lamivudine and Nevirapine, Once Daily, in Antiretroviral Naive HIV-1 Infected Patients
Brief Title: Zidovudine / Lamivudine + Nevirapine Twice Daily, Versus Tenofovir + Lamivudine + Nevirapine Once Daily in ARV-Naive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MEDEX (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAUFIN
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Hiv Infection With Antiretroviral Therapy Indication; CD4 Below 350/µL or Below 15%
Keywords: Antiretroviral Therapy; Nevirapine; HIV Viral Load; Adherence; Quality of Life; Resistance Mutations
MeSH Terms: interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
The study will compare the immuno-virological efficacy, and safety, of a once daily antiretroviral combination (tenofovir + lamivudine + nevirapine) versus a twice daily association (fixed dose combination of zidovudine/lamivudine + nevirapine) in ARV-Naive HIV-1 infected subjects, with CD4 cell count below 350/µL or below 15%, whatever the viral load. Pharmacological (nevirapine concentrations) and virologic data (resistance mutations in case of failure) will also be provided, as well as adherence rate and quality of life in respect of the treatment arms.

DETAILED DESCRIPTION:
96-week antiviral efficacy of tenofovir + lamivudine + nevirapine, once daily, versus a reference antiretroviral treatment given twice daily (zidovudine/lamivudine + nevirapine)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, confirmed by a western-blot assay, at least 6 months after primary infection
* Age > or equal to 18 years of age
* No prior antiretroviral treatment
* Karnofsky superior to 60%
* CD4 T cells < 350/µL (2 measures, with at least a 1-month interval) in women, study will be proposed when CD4 cell count is below 250/µL, as nevirapine liver toxicity increases (X10) when CD4 are > 250/µL
* Written informed consent

Exclusion Criteria:

* HIV-2 infection or co-infection
* Prior antiretroviral treatment
* Intolerance, or contraindication to investigational drugs
* Pregnant or breast-feeding woman, or plan to become pregnant
* Active untreated opportunistic infections (AIDS-defining illness, category C, CDC, 1993), or malignancies requiring cytotoxic chemotherapy
* Biological criteria: hemoglobin < 10 G/DL, neutrophil count < 1000/µL, platelets < 50000/µL, creatinine > 2N, ASAT or ALAT > 2.5N, bilirubin > 2N, hypophosphatemia
* Prevision of poor adherence
* HBC co-infection (Ag Hbs positive) or HVC co-infection (positive HCV PCR)
* Liver failure, alcohol abuse
* Treatment administration not recommended with investigational drugs
* Interferon, interleukin, or HIV vaccine treatment
* Informed consent not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-04; Study Completion 2008-06

PRIMARY OUTCOMES:
To compare the antiviral efficacy of AZT, 3TC, and NVP combination, in two doses per day, to the association of TDF, 3TC, and NVP, once a day, in antiretroviral naive HIV-1-infected patients (plasma viral load below 400 copies/ml at 96 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: REY MR DAVID, M.D, Principal Investigator — CISIH CHRU STRASBOURG
Locations (1):
- Cisih, Clinique Medical A, Hopitaux Universitaires, Strasbourg, Alsace, France